CLINICAL TRIAL: NCT04741152
Title: Blinded Resection Avoided in Case of the Pancreatic Insulinoma
Brief Title: Blinded Resection in Case of the Pancreatic Insulinoma
Status: Completed | Type: Observational
Sponsor: Vishnevsky Center of Surgery (Other)
Responsible Party: Principal Investigator, Ayrat Kaldarov, Dr. Ayrat Kaldarov, Vishnevsky Center of Surgery
Other Study IDs: 1899898189bf
Record Dates: First submitted 2021-02-04; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Insulinoma; Pancreas
Keywords: Insulinoma; Hypoglicemia; Blind resection; Hidden Insulinoma; ASVS
MeSH Terms: conditions — Insulinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Revealed insulinoma: Cases when the tumor was revealed by the preoperative diagnostics and confirmed after the tumor elimination
  Interventions: Procedure: Pancreatic resection
- Hidden Insulioma: Group when the insulinoma haven't been revealed preoperative and intraoperatively and the blind resection was performed.
  Interventions: Procedure: Pancreatic resection

INTERVENTIONS:
Procedure: Pancreatic resection — Different pancreatic resections

SUMMARY:
The blinded resection avoided in case of pancreatic insulinoma

DETAILED DESCRIPTION:
Despite of the technique and technology developement there are still a lot of troubles to verify small benign-looking pancreatic NETs. It can be especially important in case of insulinoma. The organic hyperilsulinism and severe hypoglicemia causeb by the insulin/proinsulin - producing lesion can lead to severe complications and evem death.

There are some cases of the blinded resections of the pancreas in patients with the "hidden" insulinoma when the tumor can't be revealed during the preoperative diagnostics and intraoperatively. Unfortunately, blind resection do not solve the problem of the hypoglicemia but also cause the specific pancreatic complications.

ELIGIBILITY:
Inclusion Criteria:

The blinded resection of the insulinoma

Exclusion Criteria:

Other tumors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients surgically treated in case of pancreatic insulinoma/proinsulinoma
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
No hidden insulinomas | 2010 June - 2020 June
  To improve the diagnostics of the tumor before and during the surgery. The "hidden" insulinomas haven't been diagnosed. The frozen section have to be routinely performed. The surgery haven't been finished before the morphologic confirmation of the resected lesion.

IPD SHARING:
Plan to Share IPD: No